CLINICAL TRIAL: NCT06511882
Title: Discontinuation of Hypomethylating Agent and Venetoclax in Patients With Newly Diagnosed Acute Myeloid Leukemia (AML) Who Have Achieved Negative Measurable Residual Disease (MRD)
Brief Title: Discontinuation of Hypomethylating Agent and Venetoclax in Patients With AML MRD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22191
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Decitabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Consolidation and Discontinuation (Other): Consolidation: Patient will receive HMA (azacitidine or decitabine)/VEN (venetoclax) as part of standard of care treatment.
  At the conclusion of consolidation, if the results of the bone marrow biopsy are a negative Measurable Residual Disease (MRD), patient will continue to Discontinuation.
  Discontinuation:
  Monthly clinic visits with laboratory assessment and bone marrow biopsies (BMBs) with MRD testing every 3 months to closely monitor disease status. At any point of the study if molecular relapse (including MRD emergence), or morphologic relapse, therapy will be reinitiated.
  If only molecular relapse, HMA (azacitidine or decitabine)/VEN (venetoclax) will be reinitiated with the same monitoring schedule as before.
  If morphologic relapse, HMA (azacitidine or decitabine)/VEN (venetoclax) will be reinitiated for 2 cycles.
  If no response (NR), patient will be taken off Study.
  Interventions: Drug: Azacitidine; Drug: Decitabine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Standard of Care Intravenous (IV) infusion
  Other Names: Vidaza
Drug: Decitabine — Standard of Care Intravenous (IV) infusion
  Other Names: DACOGEN
Drug: Venetoclax — Standard of Care PO (By Mouth)
  Other Names: Venclexta

SUMMARY:
The purpose of this research study is to see if people whose Acute myeloid leukemia (AML) is being successfully treated with azacitidine or decitabine in combination with venetoclax can discontinue this chemotherapy for some period of time after a year of treatment without increasing the likelihood that their AML will return.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older at the time of obtaining informed consent.
* Diagnosed with Acute Myeloid Leukemia (AML) (non-M3) as defined by 2016 World Health Organization (WHO)
* Eastern Cooperative Group (ECOG) performance status score ≤ 2
* Currently on frontline therapy with HMA (azacitidine or decitabine)/VEN and achieved Complete Remission (CR)/Complete Remission with incomplete marrow recovery (CRi) with MRD negativity defined as < 0.1% by Multiparameter Flow Cytometry (MFC)
* Within 12 months of starting HMA (azacitidine or decitabine)/VEN
* Ineligible for or declined allogeneic hematopoietic cell transplantation (HCT)
* Ability to understand and the willingness to sign a written informed consent document
* Must agree to adhere to the study visit schedule and other protocol requirements
* Patients must be able to provide adequate Bone Marrow (BM) aspirate and biopsy specimens for histopathological and Measurable Residual Disease analysis during the screening procedure

Exclusion Criteria:

* Use of cytotoxic chemotherapeutic agents, or experimental agents (agents that are not commercially available) for the treatment of AML within 28 days, or 5 half-lives, at the start of the study. Only patients who are receiving frontline HMA (azacitidine or decitabine)/VEN are potentially eligible, but if they had received a course of hydroxyurea prior to achieving CR/CRi, this is allowed.
* Any serious medical condition or uncontrolled current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or will place the subject at unacceptable risk if he/she participates in the study. Controlled infections or other medical conditions on long-term therapy is allowed.
* Patients who harbored TP53 mutation at diagnosis
* AML with extramedullary involvement including central nervous system (CNS) involvement, myeloid sarcoma, and leukemia cutis requiring directed therapy at the time of enrollment.
* Patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Rates of Complete Response (CR)/Complete Response with incomplete hematologic recovery (CRi) | Up to 18 Months
  Rates of CR/CRi at 18 months from the time of initial CR/CRi in patients who discontinue frontline HMA (azacitidine or decitabine)/VEN (venetoclax) after achieving Measurable Residual Disease (MRD) negativity by MFC within 12 months of starting therapy.
  The Null hypothesis (p0) will be tested against the alternative hypothesis (p1).
  Null hypothesis: p0 ≤ 50% will remain in CR/CRi at 18 months from the time of initial CR/CRi Alternative hypothesis: p1 ≥ 70% will remain in CR/CRi at 18 months from the time of initial CR/CRi

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 36 Months
  Overall survival will be assessed in MRD-negative patients who discontinue HMA (azacitidine or decitabine)/VEN (venetoclx).
  Overall Survival (OS) is defined as the length of time from the start of treatment until death due to any cause.
Rates to Re-Treatment | Up to 36 Months
  Rates to re-treatment is defined as Measurable Residual Disease (MRD)-negative CR/CRi and CR/CRi and rates to re-treatment following molecular or morphologic relapse duration discontinuation.
Treatment Free Molecular Remission (TFMR) | Up to 36 Months
  Defined as time from Measurable Residual Disease (MRD) negativity to first MRD positivity
European Organization for Research and Treatment of Cancer (EORTC-QLQ-C30)/Quality of Life (QoL) | Day 1 (start of enrollment), start of Discontinuation Phase, and monthly until EOT (Up to 36 Months)
  EORTC-QLQ-C30/QoL consists of a 30-item subject self-report questionnaire composed of five functional scales (physical, role, emotional, social, and cognitive), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status/quality of life scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).
  Scale scores range from 0-100.
Patient Reported Outcome Measurement Information System (PROMIS) | Day 1 (start of enrollment), start of Discontinuation Phase, and monthly until EOT (Up to 36 Months)
  PROMIS scale provides response options 1-5 to indicate patient-reported health status measures for physical, mental, and social well-being.
  It measures concepts such as pain, fatigue, physical function, depression, anxiety, and social function.
EuroQoL-5 Dimensions-5 Levels (EQ-5D-5L) Visual Analog Scale (VAS) | Day 1 (start of enrollment), start of Discontinuation Phase, and monthly until EOT (Up to 36 Months)
  EQ-5D-5L VAS is an instrument for measuring the general health status of an individual. It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Scale scores range from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Onyee Chan, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/